CLINICAL TRIAL: NCT00548249
Title: A Dose Ranging Study of Dialysate Containing Soluble Ferric Pyrophosphate (SFP) Versus Control in Subjects With ESRD Receiving Chronic Hemodialysis.
Brief Title: Dose Ranging Study of Dialysate Containing Soluble Iron to Treat Subjects With End Stage Renal Disease (ESRD) Receiving Chronic Hemodialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rockwell Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RMTI-SFP-2
Record Dates: First submitted 2007-10-19; First posted 2007-10-23 (Estimated); Results first posted 2011-02-08 (Estimated); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: End-Stage Renal Disease (ESRD)
Keywords: Subjects with ESRD receiving chronic Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — spleen fibrinolytic proteinase (human)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 0 µg iron/dL of dialysate (Placebo Comparator): Placebo 0 micrograms (µg) of iron/ deciliter (dL) of dialysate
  Interventions: Device: Standard Bicarbonate Solution
- 5 µg iron/dL of dialysate (Experimental): 5 micrograms (µg) of iron/ deciliter (dL) of dialysate
  Interventions: Drug: Soluble Ferric Pyrophosphate
- 10 µg iron/dL of dialysate (Experimental): 10 micrograms (µg) of iron/ deciliter (dL) of dialysate
  Interventions: Drug: Soluble Ferric Pyrophosphate
- 12 µg iron/dL of dialysate (Experimental): 12 micrograms (µg) of iron/ deciliter (dL) of dialysate
  Interventions: Drug: Soluble Ferric Pyrophosphate
- 15 µg iron/dL of dialysate (Experimental): 15 micrograms (µg) of iron/ deciliter (dL) of dialysate
  Interventions: Drug: Soluble Ferric Pyrophosphate

INTERVENTIONS:
Device: Standard Bicarbonate Solution — Patients received 0 micrograms (µg) of iron/ decilited (dL) of dialysate during dialysis 3 times/week for up to 26 weeks.
  Other Names: Placebo
  Arms: 0 µg iron/dL of dialysate
Drug: Soluble Ferric Pyrophosphate — Patients received 5 micrograms (µg) of iron/ decilited (dL) of dialysate during dialysis 3 times/week for up to 26 weeks.
  Other Names: SFP
  Arms: 5 µg iron/dL of dialysate
Drug: Soluble Ferric Pyrophosphate — Patients received 10 micrograms (µg) of iron/ decilited (dL) of dialysate during dialysis 3 times/week for up to 26 weeks.
  Other Names: SFP
  Arms: 10 µg iron/dL of dialysate
Drug: Soluble Ferric Pyrophosphate — Patients received 12 micrograms (µg) of iron/ decilited (dL) of dialysate during dialysis 3 times/week for up to 26 weeks.
  Other Names: SFP
  Arms: 12 µg iron/dL of dialysate
Drug: Soluble Ferric Pyrophosphate — Patients received 15 micrograms (µg) of iron/ decilited (dL) of dialysate during dialysis 3 times/week for up to 26 weeks.
  Other Names: SFP
  Arms: 15 µg iron/dL of dialysate

SUMMARY:
The purpose of this study is to determine whether Dialysate containing soluble iron (Soluble Ferric Pyrophosphate) is safe and effective in maintaining physiological iron levels during chronic hemodialysis.

DETAILED DESCRIPTION:
The study was designed to evaluate the efficacy of SFP-containing dialysate solution in maintaining physiological iron levels during chronic hemodialysis, as measured by the primary endpoint of the percent of patients whose Hemoglobin (Hgb) decreased by at least 1.0 gram/ deciliter (g/dL) from baseline. The efficacy and safety findings are to be used to determine the optimal concentration of SFP needed to safely maintain iron levels, compensating for iron losses during chronic hemodialysis.

ELIGIBILITY:
Selected Inclusion Criteria:

1. Adult subject ≥ 18 years of age undergoing chronic hemodialysis for end-stage renal disease (ESRD) three times a week
2. Hemoglobin (Hgb) values on two successive screening/baseline measures immediately prior to the start of the study averaging 10.1 to 11.5 grams/ deciliter (g/dL), inclusive
3. Transferrin Saturation (TSAT) values that average 20% or more, but not exceeding 35%, prior to dialysis measured during the screening period
4. Ferritin values that average 200 to 800 micrograms/ liter (µg/L), inclusive, measured during the screening period. An average ferritin above 800 µg/L but no greater than 1200 µg/L is allowed if the average TSAT is 20% to no greater than 25%.
5. Except for vascular access surgery, subject has no hospitalization in previous three months for a significant illness that, in the opinion of the Investigator, confers a significant risk of hospitalization during the course of the study. No blood transfusions within the last 4 weeks are allowed.
6. Subject has an adequate dialyzer blood flow rate that is acceptable to the Principal Investigator

Exclusion Criteria:

1. Hemoglobin (Hgb) values on two successive baseline/screening measurements that average ≥ 11.6g/dL
2. Subject with a current malignancy involving a site other than skin
3. Subject with a history of drug or alcohol abuse within the last six months
4. Subject believed to be unable to complete the entire study (e.g., due to a concurrent disease, life expectancy of less than a year)
5. Subject who the Principal Investigator considers will be placed at increased risk by the study procedures
6. Subject requiring hemodialysis more than 3 times per week on a regular basis.
7. Subject who is unable to discontinue oral iron or intravenous iron supplements for the duration of the study
8. Subject who is pregnant
9. Subject considered incompetent to give an informed consent
10. Subject with a positive test for Hepatitis B Surface Antigen within the past 30 days or during screening
11. Subject with known HIV infection (if this is not known, no HIV testing will be performed)
12. Subject with cirrhosis of the liver based on histological criteria or clinical criteria (presence of ascites, esophageal varices, spider nevi, or history of hepatic encephalopathy). Subject with hepatitis C, in the absence of cirrhosis, is not excluded from participation in the study if ALT and AST levels are below 2 times the upper limit of normal consistently during the 2 months preceding enrollment
13. Subject with active tuberculosis, fungal, viral, or parasitic infection
14. Subject with active bacterial infection requiring antibiotic therapy
15. Subject with pre-dialysis Corrected Q-wave to T-wave (QTc) interval ≥ 470 milliseconds (ms)
16. Subject with a history of hypokalemia, decompensated heart failure, or family history of Long QT Syndrome that in the Investigator's judgment poses a risk for Torsades de Pointe during the study
17. Subject using concomitant medications known to prolong QT/QTc interval (See Appendix I, TABLE A)
18. Subject receiving more than 60,000 units or 120 micrograms of erythropoietin (Epogen®, Procrit®, or Aranesp®) per week
19. Subject has participated in another clinical trial within 30 days of signing Informed Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2007-08; Primary Completion 2009-10 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Yocum, MD, Study Director — Rockwell Medical Technologies
Locations (28):
- United States (27):
  - Investigator, Tempe, Arizona
  - Investigator, Hacienda Heights, California
  - Investigator, Los Angeles, California
  - Investigator, Whittier, California
  - Investigative Site, Augusta, Georgia
  - Investigator, Meridian, Idaho
  - Investigator, Chicago, Illinois
  - Investigative Site, Louisville, Kentucky
  - Investigator, New Orleans, Louisiana
  - Investigator, Springfield, Massachusetts
  - Investigative Site, Detroit, Michigan
  - Investigator, Hackensack, New Jersey
  - Investigator, Brooklyn, New York
  - Investigator, Great Neck, New York
  - Investigator, Mineola, New York
  - Investigator, New York, New York
  - Investigator, Ridgewood, New York
  - Investigator, Winston-Salem, North Carolina
  - Investigative Site, Canton, Ohio
  - Investigator, Cincinnati, Ohio
  - Investigative Site, Hershey, Pennsylvania
  - Investigator, Arlington, Texas
  - Investigator, Fort Worth, Texas
  - Investigator, McAllen, Texas
  - Investigator, San Antonio, Texas
  - Investigator, Arlington, Virginia
  - Investigator, Seattle, Washington
- Investigative Site, Edmonton, Alberta, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 131 patients randomized and dosed between 27 Aug 2007 and 28 Apr 2009, across 29 study sites in U.S. and Canada.
Pre-assignment Details: No run-in or transition.
Groups:
- 0 µg Iron/dL of Dialysate: Placebo; 0 micrograms (µg) iron/deciliter (dL) of dialysate during dialysis 3 times/ week
- 5 µg Iron/dL of Dialysate: 5 micrograms (µg) iron/deciliter (dL) of dialysate during dialysis 3 times/ week
- 10 µg Iron/dL of Dialysate: 10 micrograms (µg) iron/deciliter (dL) of dialysate during dialysis 3 times/ week
- 12 µg Iron/dL of Dialysate: 12 micrograms (µg) iron/deciliter (dL) of dialysate during dialysis 3 times/ week
- 15 µg Iron/dL of Dialysate: 15 micrograms (µg) iron/deciliter (dL) of dialysate during dialysis 3 times/ week
Period: Overall Study
Arm/Group | 0 µg Iron/dL of Dialysate | 5 µg Iron/dL of Dialysate | 10 µg Iron/dL of Dialysate | 12 µg Iron/dL of Dialysate | 15 µg Iron/dL of Dialysate
Started | 26 | 26 | 29 | 22 | 28
Completed | 10 | 13 | 9 | 9 | 7
Not Completed | 16 | 13 | 20 | 13 | 21
Not completed — Hemoglobin (Hgb) decrease >=1.0 g/dL | 3 | 4 | 4 | 2 | 4
Not completed — Transferrin Saturation (TSAT) <20% | 5 | 1 | 3 | 1 | 2
Not completed — Protocol Violation | 1 | 1 | 4 | 0 | 3
Not completed — Miscellaneous | 2 | 3 | 2 | 0 | 2
Not completed — Pre-dialysis (Pre-HD) TSAT >=50% | 0 | 0 | 2 | 1 | 4
Not completed — Adverse Event | 2 | 2 | 0 | 1 | 1
Not completed — Post-dialysis high TSAT or low UIBC | 0 | 0 | 1 | 3 | 2
Not completed — Erythropoietin (ESA)Dose Change Required | 0 | 0 | 1 | 2 | 2
Not completed — Hemoglobin (Hgb) >= 12.6 g/dL | 1 | 1 | 1 | 1 | 0
Not completed — Prolonged hospitalization | 0 | 0 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0
Not completed — Corrected Q-wave T-wave (QTc) increase | 0 | 1 | 0 | 0 | 1
Not completed — Sponsor's request | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0 µg Iron/dL of Dialysate | 5 µg Iron/dL of Dialysate | 10 µg Iron/dL of Dialysate | 12 µg Iron/dL of Dialysate | 15 µg Iron/dL of Dialysate | Total
Number analyzed (Participants) | 26 | 26 | 29 | 22 | 28 | 131
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 19 | 19 | 15 | 14 | 87
  >=65 years | 6 | 7 | 10 | 7 | 14 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (10.68) | 57.3 (15.48) | 57.3 (13.97) | 57.9 (12.79) | 59.8 (16.96) | 58 (14.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 13 | 7 | 11 | 50
  Male | 18 | 15 | 16 | 15 | 17 | 81
Region of Enrollment [Number; unit: participants]
  United States | 22 | 24 | 25 | 21 | 25 | 117
  Canada | 4 | 2 | 4 | 1 | 3 | 14

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects Whose Hemoglobin (Hgb) Decreases by a Total of 1.0 Grams/ Deciliter (g/dL) (or More) From Baseline on Each of Two Successive Measurements.
Description: Efficacy of a Soluble Ferric Pyrophosphate (SFP)-containing dialysate solution in maintaining physiological iron levels during chronic HD, as measured by the percent of subjects whose hgb decreases by a total of 1.0 g/dL (or more) from baseline on each of two successive measurements. Hemoglobin was obtained weekly at the mid-week dialysis treatments and compared to baseline value (average of two hgb measurements obtained at the two consecutive baseline visits prior to randomization).
Time Frame: up to 26 weeks
Population: Modified intent-to-treat population, consisting of all subjects who received any amount of randomized study medication
Measure: Number; unit: Percent of subjects
Arm/Group | 0 µg Iron/dL of Dialysate | 5 µg Iron/dL of Dialysate | 10 µg Iron/dL of Dialysate | 12 µg Iron/dL of Dialysate | 15 µg Iron/dL of Dialysate
Number analyzed (Participants) | 26 | 26 | 29 | 22 | 28
Percent of subjects | 5 | 6 [0.30 to 3.32] | 5 [0.33 to 4.09] | 4 [0.21 to 3.02] | 10 [0.60 to 5.19]
Statistical Analysis 1: Comparison: 0 µg Iron/dL of Dialysate vs 5 µg Iron/dL of Dialysate; Hazard ratio with 95% confidence intervals comparing each SFP treatment group to placebo, and p-value from cox proportional hazards model; Test type: Superiority or Other; p = 0.999, Log Rank — p-value not adjusted for multiple comparisons; Cox Proportional Hazard = 1.00, 95% CI 2-sided [0.30 to 3.32]
Statistical Analysis 2: Comparison: 0 µg Iron/dL of Dialysate vs 10 µg Iron/dL of Dialysate; Test type: Superiority or Other; p = 0.807, Log Rank; Cox Proportional Hazard = 1.17, 95% CI 2-sided [0.33 to 4.09]
Statistical Analysis 3: Comparison: 0 µg Iron/dL of Dialysate vs 12 µg Iron/dL of Dialysate; Test type: Superiority or Other; p = 0.748, Log Rank; Cox Proportional Hazard = 0.80, 95% CI 2-sided [0.21 to 3.02]
Statistical Analysis 4: Comparison: 0 µg Iron/dL of Dialysate vs 15 µg Iron/dL of Dialysate; Test type: Superiority or Other; p = 0.299, Log Rank; Cox Proportional Hazard = 1.77, 95% CI 2-sided [0.60 to 5.19]

2. Secondary Outcome: Change From Baseline in Hemoglobin (Hgb)
Time Frame: two time points: baseline and final evaluation (last post baseline assessment, up to 26 weeks)
Population: Modified intent-to-treat population, consisting of all subjects who received any amount of randomized study medication
Measure: Mean (Standard Deviation); unit: grams/ deciliter (g/dL)
Arm/Group | 0 µg Iron/dL of Dialysate | 5 µg Iron/dL of Dialysate | 10 µg Iron/dL of Dialysate | 12 µg Iron/dL of Dialysate | 15 µg Iron/dL of Dialysate
Number analyzed (Participants) | 26 | 26 | 29 | 22 | 28
grams/ deciliter (g/dL) | -0.177 (1.1151) | 0.258 (1.4643) | 0.462 (1.2214) | 0.173 (1.5806) | -0.018 (1.2532)
Statistical Analysis 1: Comparison: 0 µg Iron/dL of Dialysate vs 5 µg Iron/dL of Dialysate; Each dose was compared to placebo using an ANOVA model with treatment as the effect; Test type: Superiority or Other; p = 0.234, ANOVA — Threshold for statistical significance p < 0.05
Statistical Analysis 2: Comparison: 0 µg Iron/dL of Dialysate vs 10 µg Iron/dL of Dialysate; Each dose was compared to placebo using an ANOVA model with treatment as the effect; Test type: Superiority or Other; p = 0.049, ANOVA — Threshold for statistical significance p < 0.05
Statistical Analysis 3: Comparison: 0 µg Iron/dL of Dialysate vs 12 µg Iron/dL of Dialysate; Each dose was compared to placebo using an ANOVA model with treatment as the effect; Test type: Superiority or Other; p = 0.375, ANOVA — Threshold for statistical significance p < 0.05
Statistical Analysis 4: Comparison: 0 µg Iron/dL of Dialysate vs 15 µg Iron/dL of Dialysate; Each dose was compared to placebo using an ANOVA model with treatment as the effect; Test type: Superiority or Other; p = 0.625, ANOVA — Threshold for statistical significance p < 0.05

3. Secondary Outcome: Time in Days for Hgb to Decrease by a Total of > = 1.0 g/dL From Baseline on Each of Two Successive Measurements in Each Treatment Group.
Description: Kaplan-Meier Estimate of Time to First Hgb Decrease by >= 1.0 g/dL
Time Frame: Up to 26 weeks
Population: Modified intent-to-treat population, consisting of all subjects who received any amount of randomized study medication.
  Because of the small number of patients reaching the endpoint of decrease in Hgb >= 1.0 g/dL, the Kaplan-Meier analysis could not estimate the number of days for at least one treatment group for the 50th percentile and higher.
Measure: Number; unit: Days
Arm/Group | 0 µg Iron/dL of Dialysate | 5 µg Iron/dL of Dialysate | 10 µg Iron/dL of Dialysate | 12 µg Iron/dL of Dialysate | 15 µg Iron/dL of Dialysate
Number analyzed (Participants) | 26 | 26 | 29 | 22 | 28
Days
  5th Percentile | 59 (0.3267) | 24 (0.6674) | 10 (0.4402) | 31 (0.3697) | 31 (0.6609)
  10th Percentile | 94 | 31 | 106 | 45 | 31
  15th Percentile | 94 | 66 | 106 | 115 | 38
  20th Percentile | 115 | 87 | 106 | 115 | 80
  25th Percentile | 115 | 108 | 115 | 150 | 94

4. Secondary Outcome: Reticulocyte Hemoglobin (CHr) Values Every Four Weeks, and at the End of the Subject's Treatment.
Description: Efficacy of SFP administration in dialysate solution as measured by Chr values every four weeks, and at the end of the Subject's Treatment (up to 26 weeks).
Time Frame: Every 4 weeks
Population: Modified intent-to-treat population, consisting of all subjects who received any amount of randomized study medication
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | 0 µg Iron/dL of Dialysate | 5 µg Iron/dL of Dialysate | 10 µg Iron/dL of Dialysate | 12 µg Iron/dL of Dialysate | 15 µg Iron/dL of Dialysate
Number analyzed (Participants) | 26 | 26 | 29 | 22 | 28
pg
  Baseline Reticulocyte Hemoglobin | 32.55 (2.084) | 32.98 (1.763) | 32.86 (3.192) | 32.34 (2.975) | 32.64 (1.858)
  Reticulocyte Hemoglobin/ Week 1 | 32.42 (2.852) | 32.58 (1.932) | 32.69 (3.019) | 31.87 (2.963) | 32.40 (2.006)
  Reticulocyte Hemoglobin/ Week 4 | 32.00 (2.668) | 32.27 (2.090) | 32.69 (2.931) | 31.82 (2.515) | 32.05 (1.837)
  Reticulocyte Hemoglobin/ Week 8 | 32.14 (2.664) | 32.28 (2.135) | 32.75 (2.985) | 31.75 (2.473) | 32.35 (1.917)
  Reticulocyte Hemoglobin/ Week 12 | 31.83 (2.347) | 32.13 (1.792) | 32.78 (1.560) | 31.82 (3.150) | 32.48 (1.894)
  Reticulocyte Hemoglobin/ Week 16 | 31.45 (2.546) | 31.95 (1.866) | 33.05 (2.396) | 31.86 (3.410) | 32.25 (2.382)
  Reticulocyte Hemoglobin/ Week 20 | 31.13 (2.172) | 31.81 (1.860) | 32.81 (2.328) | 30.68 (2.026) | 31.64 (1.338)
  Reticulocyte Hemoglobin/ Week 24 | 30.93 (2.127) | 31.85 (1.820) | 32.08 (2.680) | 30.53 (2.071) | 31.40 (1.949)
  Reticulocyte Hemoglobin/ Week 26 | 30.78 (2.638) | 31.32 (2.404) | 32.20 (2.372) | 30.72 (2.515) | 30.43 (2.600)
  Reticulocyte Hemoglobin/ End of Trial | 30.06 (1.841) | 31.50 (2.348) | 31.46 (2.352) | 30.55 (2.523) | 30.11 (2.361)
  Reticulocyte Hemoglobin/ Final Evaluation | 31.85 (2.796) | 31.68 (2.386) | 32.19 (3.026) | 31.65 (3.409) | 32.13 (2.246)

5. Secondary Outcome: Number of Subjects With Infection Episodes Requiring Antibiotic or Anti-fungal Therapy in Each Treatment Group.
Time Frame: At each dialysis session for up to 26 weeks
Measure: Number; unit: Subjects
Arm/Group | 0 µg Iron/dL of Dialysate | 5 µg Iron/dL of Dialysate | 10 µg Iron/dL of Dialysate | 12 µg Iron/dL of Dialysate | 15 µg Iron/dL of Dialysate
Number analyzed (Participants) | 26 | 26 | 29 | 22 | 28
Subjects | 2 | 1 | 2 | 0 | 1

6. Secondary Outcome: Number of Subjects With a Rise in Hemoglobin (Hgb) to 12.6 g/dL or More on Two Separate Occasions Measured One Week Apart.
Time Frame: two separate sessions measured one week apart.
Population: Modified intent-to-treat population, consisting of all subjects who received any amount of randomized study medication
Measure: Number; unit: Subjects
Arm/Group | 0 µg Iron/dL of Dialysate | 5 µg Iron/dL of Dialysate | 10 µg Iron/dL of Dialysate | 12 µg Iron/dL of Dialysate | 15 µg Iron/dL of Dialysate
Number analyzed (Participants) | 26 | 26 | 29 | 22 | 28
Subjects | 6 | 6 [0.33 to 3.17] | 9 [0.67 to 5.32] | 7 [0.48 to 4.22] | 8 [0.43 to 3.60]

ADVERSE EVENTS:
Time Frame: Up to 26 weeks
Arm/Group | 0 µg Iron/dL of Dialysate | 5 µg Iron/dL of Dialysate | 10 µg Iron/dL of Dialysate | 12 µg Iron/dL of Dialysate | 15 µg Iron/dL of Dialysate
Serious Adverse Events (participants affected / at risk) | 7/26 | 2/26 | 5/29 | 7/22 | 5/28
Other Adverse Events (participants affected / at risk) | 20/26 | 17/26 | 20/29 | 16/22 | 17/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0 µg Iron/dL of Dialysate (N=26) | 5 µg Iron/dL of Dialysate (N=26) | 10 µg Iron/dL of Dialysate (N=29) | 12 µg Iron/dL of Dialysate (N=22) | 15 µg Iron/dL of Dialysate (N=28)
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 1 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Catheter bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Thalamic infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Chronic obstructive pulmonary (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypertensive emergency (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Graft dysfunction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0 µg Iron/dL of Dialysate (N=26) | 5 µg Iron/dL of Dialysate (N=26) | 10 µg Iron/dL of Dialysate (N=29) | 12 µg Iron/dL of Dialysate (N=22) | 15 µg Iron/dL of Dialysate (N=28)
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 7 | 2 | 4
Nausea (Gastrointestinal disorders) | 4 | 3 | 2 | 6 | 4
Vomiting (Gastrointestinal disorders) | 3 | 3 | 2 | 4 | 1
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 3 | 0 | 2 | 1
Oedema peripheral (General disorders) | 5 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 2 | 0 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 1 | 1
Asthenia (General disorders) | 2 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 2 | 0
Feeling hot (General disorders) | 0 | 1 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 3 | 1
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 1 | 2
Bronchitis (Infections and infestations) | 0 | 2 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 3 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 2 | 4 | 5 | 2 | 4
Thrombosis in device (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2 | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1 | 1
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 1
Contusion (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Procedural hypertension (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Serum ferritin increased (Investigations) | 1 | 0 | 1 | 0 | 1
Blood iron decreased (Investigations) | 0 | 1 | 0 | 0 | 1
Iron binding capacity unsaturated decreased (Investigations) | 0 | 1 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 0 | 4 | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 5 | 2 | 5 | 3 | 2
Dizziness (Nervous system disorders) | 2 | 3 | 4 | 1 | 2
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3 | 4 | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
AE tabulation best summarizes the primary safety outcome.

Lack of accuracy in analytical method for measuring iron concentration in inflow and outflow from dialysis machine impaired ability to assess secondary outcome of amount SFP transferred.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No